CLINICAL TRIAL: NCT03703752
Title: CT Images and Clinical Relevance of Internal Hernia
Brief Title: CT and Clinical Features of Internal Hernia
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Lei Dou, principal investigator, Tongji Hospital
Other Study IDs: TJ-10207102
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: CT Images of Internal Hernia; Clinical Outcomes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adhesive IH: Adhesive IH can further be divided into primary or secondary groups according to the history of abdominal and(or) pelvic surgery
  Interventions: Diagnostic Test: Multi-detector CT scan
- non-adhesive IH: Non-adhesive IH means the IH resulting from the abnormality of peritoneal structure.
  Interventions: Diagnostic Test: Multi-detector CT scan

INTERVENTIONS:
Diagnostic Test: Multi-detector CT scan — This is a diagnostic radiological test to diagnose the IH and evaluate the clinical condition of IH

SUMMARY:
Researchers retrospectively reviewed patients with internal hernia that confirmed by surgical exploration between Feb. 2012 and Feb. 2018. and analysis the Medical records and MDCT images to investigate the clinical and radiological features of internal hernia.

DETAILED DESCRIPTION:
51 Patients with definite diagnosis of IH during surgical exploration from Feb. 2012 to Feb. 2018 in our hospital were included in this research. Medical records including MDCT images and intra-operative findings were collected retrospectively. The CT features of different subgroups were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* IH confirmed by surgical exploration

Exclusion Criteria:

* diaphragmatic hernia and traumatic IH

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Patients with definite diagnosis of IH during surgical exploration from Feb. 2012 to Feb. 2018 in our hospital were included in this research
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
CT features | 2 weeks
  MDCT features of IH were assessed for the following findings: (1) Demonstration of bowels dislocation in IH: dislocated cluster of the intestinal segments; crowding or convergence of mesenteric vessels; (2) Demonstration of obstruction or ischemia: bowel wall thickening or abnormal enhancement; dilated bowels with abnormal free fluid; twisted bowels with swirl sign of vessels. (3) Demonstration of specific signs: hernial orifice and closed-loop of intestine; fat notch sign.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No